CLINICAL TRIAL: NCT07313800
Title: Enduring Migraine Benefit From Responsive Artery Coil Embolization (EMBRACE): A Single-Site, Non-Significant Risk Pilot Study of Middle Meningeal Artery Embolization Using FDA-Cleared Coils for Refractory Episodic Migraine
Brief Title: EMBRACE Study: Enduring Migraine Benefit From Responsive Artery Coil Embolization
Acronym: EMBRACE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cortex Neurovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMBRACE-001
Record Dates: First submitted 2025-12-30; First posted 2026-01-02 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Migraine Disorders; Refractory Migraine; Chronic Migraine
Keywords: Middle Meningeal Artery Embolization; MMA Embolization; Refractory Migraine; Coil Embolization; Neurovascular Intervention; Migraine Prevention; TEMMA; TEMMA procedure; TEMMA protocol; Targeted Embolization for Migraine Management
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: Single-arm, open-label pilot study evaluating outcomes following the TEMMA procedure (Targeted Embolization for Migraine Management). All enrolled participants undergo endovascular treatment targeting meningeal arterial contributors to migraine as part of the TEMMA clinical program. Adjunctive intra-procedural assessments may be performed at the discretion of the treating physician but are not required for participation and are not used as mandatory eligibility criteria. Outcomes are assessed within-subject and compared against baseline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- TEMMA Procedure (Targeted Embolization for Migraine Management) (Experimental): Participants with refractory migraine undergo the TEMMA procedure (Targeted Embolization for Migraine Management), an endovascular treatment strategy addressing meningeal arterial contributors to migraine. Treatment is performed using FDA-cleared devices per institutional clinical practice. Procedural details and adjunctive assessments are individualized and not dictated by the study protocol. Outcomes are evaluated using within-subject comparison to baseline.
  Interventions: Device: TEMMA Endovascular Treatment

INTERVENTIONS:
Device: TEMMA Endovascular Treatment — Endovascular treatment targeting meningeal arterial contributors to migraine performed as part of the TEMMA procedure (Targeted Embolization for Migraine Management) using FDA-cleared devices. Procedural techniques and adjunctive assessments are individualized at the discretion of the treating physician and are not standardized within the study.

SUMMARY:
This single-site, open-label pilot study evaluates the safety, feasibility, and potential durability of the TEMMA procedure (Targeted Embolization for Migraine Management), an endovascular treatment strategy targeting meningeal arterial contributors to migraine. Adults aged 18-60 with refractory migraine despite prior preventive therapies are eligible. The study assesses migraine outcomes over 12 months using patient-reported headache frequency, pain intensity, acute medication use, migraine-related disability (MIDAS), and quality-of-life measures (MSQ v2.1).

DETAILED DESCRIPTION:
This is an investigator-initiated, prospective, single-site, open-label pilot study designed to evaluate the safety, feasibility, and potential durability of the TEMMA procedure (Targeted Embolization for Migraine Management), an endovascular treatment approach targeting meningeal arterial contributors to migraine symptoms. TEMMA represents a structured clinical program applying endovascular treatment principles to patients with refractory migraine.

Participants undergo a baseline assessment period that includes prospective headache diary collection, capturing headache presence, pain intensity, and acute medication use, along with baseline migraine-related disability and quality-of-life assessments. Endovascular treatment is performed as part of the TEMMA program using FDA-cleared devices in accordance with institutional clinical practice. Procedural techniques, vessel selection, materials, adjunctive assessments, and treatment sequencing are determined by the treating physician and are not fully standardized within this pilot study.

Adjunctive assessments, which may include intra-procedural physiologic or pharmacologic evaluations, may be performed at the discretion of the treating physician to inform clinical decision-making but are not required for study participation and are not used as mandatory eligibility criteria.

Participants are followed longitudinally with serial headache diary data and standardized patient-reported outcome measures collected at predefined intervals through 12 months following treatment. The primary endpoint is change in monthly headache days compared with baseline. Secondary endpoints include changes in headache intensity, acute medication use, migraine-related disability, quality of life, and durability of symptom improvement.

Safety is monitored throughout the study through adverse event reporting with independent physician oversight.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* Diagnosis of migraine (with or without aura)

  -≥8 headache days per month
* Failure of ≥2 preventive medication classes
* Ability to complete electronic headache diary and surveys
* Ability to provide informed consent

Exclusion Criteria:

* Secondary headache disorders
* Prior MMA embolization
* Contraindication to angiography or embolization
* Pregnancy
* Inability to comply with follow-up

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in Monthly Headache Days Post-Embolization | Baseline to 12 months post-embolization
  Change from baseline in the number of headache days per month following bilateral middle meningeal artery coil embolization, assessed via SMS-based headache diary.

SECONDARY OUTCOMES:
Change in Headache Intensity | Baseline to 12 months post-embolization
  Change from baseline in average headache pain intensity (0-10 scale), assessed via SMS-based headache diary.
Change in Acute Medication Use | Baseline to 12 months post-embolization.
  Change from baseline in the number of days with acute migraine medication use per month.
Change in Migraine Disability Assessment (MIDAS) Score | Baseline to 3 months (assessed at 1, 3, 6, and 12 months).
  Change from baseline in MIDAS score, a validated measure of migraine-related disability.
Change in Migraine-Specific Quality of Life Questionnaire (MSQ v2.1) Score | Baseline to 3 months (assessed at 1, 3, 6, and 12 months).
  Change from baseline in MSQ v2.1 score, a validated measure of migraine-specific quality of life.
Time to Symptom Recurrence Following Lidocaine Testing | Up to 4 weeks post-lidocaine testing.
  Duration of symptom improvement (time to return to baseline headache frequency/intensity) after bilateral MMA lidocaine testing.
Time to Symptom Recurrence Following Embolization | Up to 12 months post-embolization.
  Duration of symptom improvement (time to return to baseline headache frequency/intensity) after bilateral MMA coil embolization.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Wang, MD, Principal Investigator — Cortex Neurovascular
Locations (1):
- Cortex Neurovascular / TRA Union, Tacoma, Washington, United States

IPD SHARING:
Plan to Share IPD: No